CLINICAL TRIAL: NCT05834946
Title: Identification of Biological Responses as a Causal Link for the Increased Peri-implantitis in Patients With History of Periodontitis
Brief Title: Biological Responses Affecting Early-stage Dental Implant Placement in Patients With History of Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DF RD2002/0002
Record Dates: First submitted 2023-01-17; First posted 2023-04-28 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-04

CONDITIONS: Periodontitis; Peri-implant Mucositis; Peri-Implantitis
Keywords: dental implant; history of periodontitis; matrix metalloproteinase (MMP)-8; histological analysis; next generation sequencing; dental plaque; gingival crevicular fluids; peri-implant sulcular fluids; peri-implant soft tissue; proteomic analysis
MeSH Terms: conditions — Periodontitis; Peri-Implantitis; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Test group: Patient with history of periodontitis Control group: Patient without history of periodontitis
  Patients in both groups will be randomised to receive one of two type of implants with different surface characteristics.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants will be blinded from the randomisation. An opaque envelope will be used to conceal the implant designation and will only be revealed to the operator after the site is ready for implant placement. A blinded researcher will be assigned as clinical assessor who will not be involved with the surgical procedure, subject recruitment nor consent taking. An assistant who is not involved with the research will also be asked to re-code the sample tubes to ensure blinding for data/sample analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group T-A (Experimental): 7 patients with history of periodontitis
  Interventions: Other: Megagen implant placement
- Group T-B (Experimental): 7 patients with history of periodontitis
  Interventions: Other: Biomate-Swiss implant
- Group C-A (Active Comparator): 7 patients without history of periodontitis
  Interventions: Other: Megagen implant placement
- Group C-B (Active Comparator): 8 patients without history of periodontitis
  Interventions: Other: Biomate-Swiss implant

INTERVENTIONS:
Other: Megagen implant placement — Megagen implant with sand-blasted, large-grit, acid-etched (SLA) and nano-calcium ions incorporated surface
  Arms: Group C-A; Group T-A
Other: Biomate-Swiss implant — Biomate-Swiss implant with precision dimension laser (PDL) surface
  Arms: Group C-B; Group T-B

SUMMARY:
This prospective parallel, double-blind, four-arm randomised controlled clinical study is planned to assess the difference in the level of the inflammatory biomarkers expressed following the placement of the first dental implant in patients with history of periodontitis (successfully treated) and healthy controls without the disease, during implant osseointegration period. The subjects in both groups will also be randomised to receive one of the two types of implants provided which have different surface treatment.

DETAILED DESCRIPTION:
This is a prospective, parallel, double-blind, four-arm randomised clinical control study, aims to investigate the changes of clinical parameters and pro-inflammatory biomarkers expression and the shift following the first dental implant placement in patients who have been successfully treated for periodontitis, compared with healthy control without the disease.

The main questions to answer are:

1. Why do patients with history of periodontitis are at a greater risk to develop peri-implantitis than patients without history of periodontitis?
2. Is there any difference in the microbial composition, histological and immunological reaction of the host's dental plaque, peri-implant soft tissue, gingival crevicular fluids (GCF) of adjacent teeth and peri-implant sulcular fluids (PISF) following implant placement in patients with and without a history of periodontitis? The test group will consist of subjects with stabilised periodontitis, whilst the control group will consist of healthy patients with no history of periodontitis, as identified via history taking and clinical screening. Periodontal condition will be determined based on the new 2017 periodontal classification. All participants in both groups will be randomised to receive one of two types of implants with different surface treatment.

Clinical measurement, GCF and PISF will be collected around the single implant and adjacent teeth, at the following stages (time-point):

* Baseline (pre-operative)
* After implant placement (prior to the second stage surgery)
* After implant exposure (prior to the crown restoration)
* 3-month after the implant is restored
* Soft tissue will be obtained during the first stage (baseline) and second stage implant surgery (post-operative) and analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Specific inclusion criteria for test group:

   * History of periodontitis but currently stable
   * Must have successfully completed active periodontal treatment at least 4 months prior to the commencement of study
2. Specific inclusion criteria for control group:

   * No history of periodontitis, with minimal age-related radiographic bone loss
   * Reason for losing the tooth/teeth was not due to periodontal problem
3. General inclusion criteria:

   * Medically healthy
   * Aged between 30 to 65 years old
   * Non-smoker, or quit smoking at least 12 months before study commencement
   * Good oral hygiene (full mouth plaque score (FMPS)<20%, full mouth bleeding score (FMBS)<15%)
   * Indicated for a single implant placement in the posterior region, with adjacent and contralateral natural tooth
   * Intact inter-cuspal position

Exclusion Criteria:

* Previous history of dental implant placement
* Currently pregnant or intend to be pregnant, and/or lactating mothers
* Taking long-term medicines which may affect gingival tissue and oral microbiome, e.g. antibiotics, anticoagulants, anticonvulsants, immunosuppressants and calcium channel blockers.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and male
Enrollment: 29 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Level of matrix metalloproteinase (MMP)-8 expressed in the gingival crevicular and peri-implant sulcular fluids during the early-stage of dental implant placement | From baseline (1st time-point (TP1)) to 1st stage surgery (implant placement - TP2), after 2nd stage surgery (implant exposure (TP3) and 3-months after implant crown restoration (final visit- TP4)
  To measure the absolute quantification of MMP-8 level expressed during the implant osseointegration period in all study groups via ELISA method.

SECONDARY OUTCOMES:
Shift of the microbial composition in the supragingival dental plaque, identified via 16S rRNA next generation sequencing | From baseline (1st time-point (TP1)) to 1st stage surgery (implant placement - TP2), after 2nd stage surgery (implant exposure (TP3) approximately 3 months after the 1st stage surgery) and 3-months after implant crown restoration (final visit- TP4)
  Identification and comparison of supragingival dental plaque bacteria species/genus and the shift of the bacterial composition during the early-stage of dental implant placement between study groups
Shift of proteome profiles in the gingival crevicular and peri-implant sulcular fluids during the early-stage of dental implant placement | From baseline (1st time-point (TP1)) to 1st stage surgery (implant placement - TP2), after 2nd stage surgery (implant exposure (TP3) approximately 3 months after the 1st stage surgery) and 3-months after implant crown restoration (final visit- TP4)
  To assess the protein profile and levels of expression of the pro-inflammatory cytokines in GCF and gingival tissue via liquid chromatography-electrospray ionization tandem mass spectrometry (LC-MS) proteomic analysis following osseointegration.
Histological changes in the peri-implant soft tissue before and after implant placement | Between first stage (baseline/pre) and second stage implant surgery (post-operative) at 3 months after the first surgery
  Number and co-localisation of cells with MMP-8, pro-inflammatory (M1)- and anti-inflammatory (M2)-related cytokines via hematoxylin and eosin staining, immunohistochemistry and immunofluorescence analysis
Changes in the clinical parameters during the early-stage implant placement | From baseline (1st time-point (TP1)) to 1st stage surgery (implant placement - TP2), after 2nd stage surgery (implant exposure (TP3) approximately 3 months after the 1st stage surgery) and 3-months after implant crown restoration (final visit- TP4)
  To assess intra-oral clinical parameters changes (i.e. patient-level and tooth-level mean periodontal pocket depth (mm) and clinical attachment level (mm); full mouth plaque score (%) and bleeding score (%)) following the first dental implant placement, each time-point (TP). The deeper the depth/higher the level or percentage means the worse the condition is.

CONTACTS AND LOCATIONS:
Overall Officials: Norul H Mohamad-Hassan, DDS,MCD, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Dentistry, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification. Researchers should provide a methodologically sound proposal and directed to the principal investigator by email.
Time Frame: Beginning 3 months and ending 5 years following article(s) publication.
Access Criteria: To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement.